CLINICAL TRIAL: NCT01983735
Title: A Randomized, Double-blind, Multi-center, Phase 3 Trial to Evaluate the Efficacy and Safety of a Fixed Dose Combination of Telmisartan and S-Amlodipine(TELMINUVO TAB.) Versus S-Amlodipine Monotherapy in Patients With Stage 2 Hypertension
Brief Title: Efficacy and Safety of TELMINUVO to Stage 2 Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 130HT13015
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension
Keywords: TELMINUVO Tab.; CKD-828; Hypertension; Stage 2 Hypertension; S-Amlodipine; Telmisartan
MeSH Terms: conditions — Hypertension | interventions — levamlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TELMINUVO Tab. (80/2.5mg, 80/5mg) (Experimental)
  Interventions: Drug: TELMINUVO Tab. (80/2.5mg); Drug: TELMINUVO Tab. (80/5mg)
- S-Amlodipine 2.5, 5mg (Active Comparator)
  Interventions: Drug: S-amlodipine 2.5mg; Drug: S-amlodipine 5mg

INTERVENTIONS:
Drug: TELMINUVO Tab. (80/2.5mg) — * Fixed dose combination of Telmisartan 80mg and S-amlodipine 2.5mg QD 2 weeks.
  * With the others investigation product placebo 1 tab QD 2 weeks.
  Other Names: TELMINUVO Tab.
  Arms: TELMINUVO Tab. (80/2.5mg, 80/5mg)
Drug: TELMINUVO Tab. (80/5mg) — * Fixed dose combination of Telmisartan 80mg and S-amlodipine 5mg QD 6 weeks.
  * With the others investigation product placebo 1 tab QD 6 weeks.
  Other Names: TELMINUVO Tab.
  Arms: TELMINUVO Tab. (80/2.5mg, 80/5mg)
Drug: S-amlodipine 2.5mg — * S-amlodipine 2.5mg QD 2 weeks
  * With the others investigation product placebo 1 tab QD 2 weeks.
  Other Names: Anydipine S
  Arms: S-Amlodipine 2.5, 5mg
Drug: S-amlodipine 5mg — * S-amlodipine 5mg QD 6weeks
  * With the others investigation product placebo 1 tab QD 6 weeks.
  Other Names: Anydipine S
  Arms: S-Amlodipine 2.5, 5mg

SUMMARY:
The aim of present study is to evaluate the efficacy and safety of two dose combination of Telmisartan/S-Amlodipine (80/2.5mg and 80/5mg) compared with S-Amlodipine monotherapy (2.5mg and 5mg) in patients with Stage 2 hypertension.

DETAILED DESCRIPTION:
* In patients with Stage 2 hypertension to determine the efficacy and safety of Telmisartan/S-Amlodipine (80/2.5mg and 80/5mg) or S-Amlodipine monotherapy (2.5mg and 5mg) during 8 weeks.
* This study is consist of placebo run-in period(2 weeks_single blind) and treatment period(8 weeks_double blind).

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* at the screening visit

  * antihypertensive drugs not taking: 160mmHg ≤ sitSBP < 200mmHg
  * antihypertensive drugs taking: 140mmHg ≤ sitSBP < 180mmHg
* at the randomization visit(160mmHg ≤ sitSBP < 200mmHg)
* willing and able to provide written informed consent

Exclusion Criteria:

* mean sitting DBP ≥ 120mmHg or mean sitting SBP ≥ 200mmHg at the screening visit and randomization visit
* for the past four weeks based on beginning of administration, patients took over four antihypertensive drugs
* known or suspected secondary hypertension(ex. aortic coarctation, Primary hyperaldosteronism, renal artery stenosis, pheochromocytoma)
* has severe heart disease(Heart failure NYHA functional class 3, 4), ischaemic heart diseases status need to treatment, myocardiopathy, Valve disease, arrhythmia and so on and operated Coronary angioplasty
* has cerebrovascular disease as cerebral infarction, cerebral hemorrhage within 6 months
* Type I Diabetes Mellitus, Type II Diabetes Mellitus with poor glucose control as defined by fasting glucosylated hemoglobin(HbA1c) > 8%)
* known severe or malignant retinopathy
* defined by the following laboratory parameters:

  * hepatic dysfunction(AST/ALT > UNL X 3)
  * renal dysfunction(serum creatinine > UNL X 1.5)
  * hypopotassemia(K < 3.0mmol/L) or hyperpotassemia (K>5.5 mmol/L)
* acute or chronic inflammatory status need to treatment
* need to additional antihypertensive drugs during the study
* need to concomitant medications known to affect blood pressure during the study
* history of angioedema related to ACE inhibitors or Angiotensin II Receptor Blockers
* known hypersensitivity related to either study drug
* history of drug or alcohol dependency within 6 months
* any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of investigational products(ex. gastrointestinal tract surgery such as gastrectomy, gastroenterostomy or bypass, active inflammatory bowel syndrome within 12 months prior to screening, gastric ulcers need to treatment, gastrointestinal/rectal bleeding, impaired pancreatic function such as pancreatitis, obstructions of the urinary tract or difficulty in voiding)
* administration of other study drugs within 4weeks prior to screening
* premenopausal women(last menstruation > 1year) not using adequate contraception, pregnant or breast-feeding
* history of malignancy including leukemia and lymphoma within the past 5 years
* in investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Mean Sitting Systolic Blood Pressure (MSSBP) | After 8 weeks of treatment

SECONDARY OUTCOMES:
Mean Sitting Systolic Blood Pressure (MSSBP) | After 2 weeks and 4 weeks of treatment
Mean Sitting Diastolic Blood Pressure (MSDBP) | After 2weeks, 4weeks and 8 weeks of treatment
Control Rate | After 8 weeks of treatment
  Sitting SBP<140mmHg, Sitting DBP<90mmHg
Response Rate | After 8 weeks of treatment
  Reduction of Sitting SBP≥20mmHg, Sitting DBP ≥10mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- The catholic university of Korea Seoul St. Mary's hospital, Seoul, South Korea